CLINICAL TRIAL: NCT06972108
Title: Caffeine for Oxygen Dependent Meconium Aspiration Syndrome
Brief Title: CAffeine Use in Prolonged Oxygen Use in meConium aspIration Syndrome in Neonatal Outcomes (CAPUCINO)
Acronym: CAPUCINO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00140244
Record Dates: First submitted 2025-04-21; First posted 2025-05-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Meconium Aspiration Syndrome
MeSH Terms: conditions — Meconium Aspiration Syndrome | interventions — caffeine citrate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeine arm (Experimental): Caffeine at standard doses
  Interventions: Drug: Caffeine citrate
- Placebo arm (Placebo Comparator)
  Interventions: Other: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: Caffeine citrate — Caffeine citrate loading at 10 mg/kg, followed by daily maintenance of 5 mg/kg PO
  Arms: Caffeine arm
Other: Saline (NaCl 0,9 %) (placebo) — Saline PO for loading and daily maintenance
  Arms: Placebo arm

SUMMARY:
When babies are stressed in the womb, they sometimes pass meconium in the amniotic fluid. When this happens, they may swallow the meconium-stained fluid into their lungs which may cause them to have poor oxygen levels and require resuscitation and significant breathing support in the early hours after birth. This is referred to as Meconium Aspiration Syndrome (MAS). Some babies may recover slowly and require breathing and/or oxygen support for days. Caffeine is a drug that can help improve breathing efforts and is commonly used in premature babies who do not have regular or strong breathing efforts. Caffeine has been used in babies with MAS who recovered slowly (i.e. requiring breathing or oxygen support for a longer period) for several years now. Despite having success in many babies, there is no evidence to examine its effectiveness and mechanism of action. This pilot study proposes to look at the effects of caffeine in babies with MAS who require ongoing breathing and oxygen support. There will also be examination of whether caffeine improves breathing efforts with better lung opening using ultrasound images of the lungs.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born through meconium-stained amniotic fluid, and
2. Gestational age at or greater than 35+0 weeks at birth, and
3. Postnatal age of 10 to 14 days-old, and
4. Full enteral feeds either at semi-demand with a mix of gavage or oral feeds or at full-demand feeds by oral method, and
5. Stable respiratory condition for 24-48 hours prior to enrolment, and require respiratory support defined as: receiving non-invasive respiratory support including one of the following

   1. High flow nasal cannula of less than or equal to 2L/min/Kg and FiO2 <0.25, or
   2. Low flow nasal cannula at <100 ml/min

Exclusion Criteria:

1. Preterm infants of less than 35+0 weeks gestation, or
2. Postnatal age younger than 9 day-old or older than 15 day-old, or
3. Parenteral nutrition supplementation or full enteral feeds by gavage, or
4. Received caffeine within 5 days prior to enrolment, or
5. Currently, receiving invasive respiratory support or continuous positive airway pressure (CPAP), or
6. During the study period with the administration of study medication, the infant cannot receive steroids including dexamethasone, hydrocortisone and budesonide by intravenous, enteral or inhalational route, or
7. Medical diseases including infections, electrolytes or acid-base imbalances, significant anemia, systematic and metabolic disorders that contribute to respiratory insufficiency other than meconium aspiration syndrome, or
8. Congenital anomalies including but not limited to respiratory tract malformations, congenital heart diseases, and syndromal abnormalities.

Ages: 10 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
24 hours oxygenation- 48-72 hours | 48-72 hours before the administration of caffeine or placebo
  24 hours oxygenation (SpO2) at 48-72 hours before the administration of caffeine or placebo
24 hours oxygenation - 72 hours | 72 hours after the administration of caffeine or placebo
  24 hours oxygenation (SpO2) at 72 hours after the administration of caffeine or placebo

SECONDARY OUTCOMES:
Baseline point-of-care lung ultrasound (POCUS) | At baseline
  Diaphragmatic function and lung aeration scores (0-18, 0=best and 18=worst) via POCUS at baseline
Post randomization Point-of-care lung ultrasound (POCUS) | 60-84 hours after the administration of caffeine or placebo
  Diaphragmatic function and lung aeration scores (0-18, 0=best and 18=worst) via POCUS 60-84 hours after the administration of caffeine or placebo

OTHER OUTCOMES:
Hospital Stay | Up to 10 weeks
  Duration of hospital stay
Duration of respiratory support | Up to 10 weeks
  Respiratory support during the hospital stay
Duration of oxygen therapy | Up to 10 weeks
  Oxygen therapy during the hospital stay

IPD SHARING:
Plan to Share IPD: Yes
Upon approval of the researcher group, de-identified individual participant data (IPD) collected in this study available to other researchers. IPD includes individual participant data collected throughout the course of the study and may include the analyzable data set.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Twelve months after the completion of the study
Access Criteria: The data may be obtained by direct application through the principal investigator of the study. Purpose of the use must be stated.

REFERENCES:
- [Background] Dini G, Ceccarelli S, Celi F, Semeraro CM, Gorello P, Verrotti A. Meconium aspiration syndrome: from pathophysiology to treatment. Ann Med Surg (Lond). 2024 Feb 15;86(4):2023-2031. doi: 10.1097/MS9.0000000000001835. eCollection 2024 Apr. PMID 38576961